CLINICAL TRIAL: NCT04196478
Title: Role of Color Doppler Ultrasonography in Assessment of Vascular Access Surveillance in Hemodialysis Patients.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Lina Farid, Lina Mohamed Farid, Assiut University
Other Study IDs: DUS in vascular accesses
Record Dates: First submitted 2019-12-02; First posted 2019-12-12 (Actual); Last update posted 2019-12-12 (Actual); Status verified 2019-12

CONDITIONS: Arteriovenous Fistula
MeSH Terms: conditions — Arteriovenous Fistula | interventions — Ultrasonography, Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: doppler ultrasound — a 7.5 MHz ultrasound (US) linear probe is needed, grey-scale ultrasound and Color Doppler and a minimum display facility of the Doppler velocity spectrum for blood flow calculation are mandatory tools.

SUMMARY:
The aim of this study is to provide an overview of the possible applications of DUS during the maturation and postoperative follow-up of vascular access, with particular emphasis to establish a relationship between doppler Ultrasound parameters including:

1. Flow volume.
2. Outflow vein diameter.
3. Outflow vein depth.
4. Resistive index.

ELIGIBILITY:
Inclusion Criteria:

* ESRD patients on dialysis with heamodialysis vascular access with adult age group (18 years and above).

Exclusion Criteria:

* Patients with chronically occluded vascular access with failed surgical or interventional attempts.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — adult group
Study Population: Sample size was calculated using Epi-Info 7 software. According to the results of previous study conducted at renal dialysis unit of Assiut university hospital (7) the most common complication occurred in haemodialysis access (A-V fistula) was infected A-V access (23.8%). Based on this prevalence the minimum required sample size for current study is 84 patients.
  Following assumptions were used to calculate this sample:
  Target population size = 120 (as number of new haemodialysis patients is 100-120 each year).
  N.B: in this study we will include all eligible cases at renal dialysis unit of Assiut university i.e., patients of last year (total coverage sample)
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2020-01-01 (Estimated); Primary Completion 2021-01-01 (Estimated); Study Completion 2021-01-01 (Estimated)

PRIMARY OUTCOMES:
Maturation of arteriovenous fistulas | 6 weeks duration follow up
  Assess the role of grey scale and color Doppler US in the early detection of failure in the hemodialysis vascular access.
  Maturation and monitoring\ surveillance of arteriovenous fistula.

IPD SHARING:
Plan to Share IPD: Undecided